CLINICAL TRIAL: NCT03777267
Title: Cereset Research Exploratory Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00055280
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Neurological Diseases or Conditions; Cardiovascular Conditions After Birth; Psychophysiologic Disorders
Keywords: Stress; Neurotechnology; Autonomic Dysregulation; Hyperarousal; Brain electrical activity; Allostasis; HIRREM; Cereset Research; Insomnia; Anxiety
MeSH Terms: conditions — Psychophysiologic Disorders; Primary Dysautonomias; Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This will be a single site, open label, pilot clinical trial, enrolling people aged 11 or older, who have self-reported symptoms of stress, anxiety, or insomnia, and meet a threshold score on self-reported inventories. Up to 200 participants will be enrolled so as to gather pilot data that will help inform regarding effect size, and dosing to support future cohort-specific randomized trials. Participants will receive between 4 and 12 intervention sessions of Cereset Research consisting of audible tones echoing current brainwave activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Experimental: Active CR (Experimental): For this single arm, open label, exploratory trial this will be the intervention arm using active CR.
  Interventions: Device: Active CR

INTERVENTIONS:
Device: Active CR — The upgraded platform for medical research using the HIRREM technology has been rebranded as Cereset Research® (CR). This system uses the same core technology and algorithms to echo brainwaves in real-time using audible tones, as with HIRREM. The CR system also includes 64-bit processing architecture for faster feedback, the use of 4 sensors, and the use of standard protocols (with flexibility regarding the length and sequencing of the standard protocols), all done with eyes closed. Four sensors are applied to the scalp at a time. However, only two sensors are actively echoing feedback. The software automatically switches from one sensor pair to the other when needed. This reduces the number of sensor placement changes needed, resulting in shorter session time and fewer interruptions.

SUMMARY:
The purpose of this study is to evaluate the use of Cereset Research to improve autonomic function in participants with symptoms of stress, anxiety, or insomnia.

DETAILED DESCRIPTION:
The primary objective of this open label exploratory study is to evaluate the effect of CR to improve autonomic cardiovascular regulation in participants with symptoms of stress, anxiety, or insomnia.

The secondary objective is to evaluate the effect of CR on a variety of self-reported symptom inventories.

Tertiary objectives are to explore the impact of selected medications on outcomes associated with use of CR, the effect size in subgroups of participants who also report specific co-morbid symptoms or conditions of interest, and any unexpected challenges or barriers for working with the same. The latter includes those with TBI, PTSD, hypertension, hot flashes, chronic pain, or prior stroke.

Methods: This will be a single site, open label, pilot clinical trial, enrolling people aged 11 or older, who have self-reported symptoms of stress, anxiety, or insomnia, and meet a threshold score on self-reported inventories. Up to 200 participants will be enrolled. Participants will receive between 4 and 12 sessions of audible tones echoing current brainwave activity (CR). Participants will continue their other current care throughout the study. There will be pre- and post-intervention data collection of physiological outcomes (BP, HR, and measures of autonomic cardiovascular regulation assessed by heart rate variability and baroreflex sensitivity), which will also serve as the primary outcome. Secondary outcomes to be collected include symptom inventories for insomnia (Insomnia Severity Index, ISI; depression (Center for Epidemiological Studies- Depression Scale, CES-D), anxiety (Generalized Anxiety Disorder-7, GAD-7), and stress (Perceived Stress Scale, PSS). Other tertiary measures include traumatic stress (PTSD Checklist for civilians, PCL-C, or military, PCL-M), and overall quality of life (QOLS). Participants who also self-report having specific co-morbid symptoms or conditions of interest may complete additional condition-specific outcome measures. All measures will be collected at an enrollment visit (V1), and the intervention will begin 0-14 days thereafter. Mean contrasts will be used to compare the changes in measures of autonomic cardiovascular regulation from V1 to V3, the primary outcome, as well as for secondary and appropriate tertiary outcomes. Linear mixed models, which can accommodate within-subject correlations due to repeated assessments over time, will be used to generate point estimates for effect size along with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have the ability to comply with basic instructions and be able to sit still comfortably with the sensor leads attached
* Subjects experiencing symptoms of stress, anxiety, or insomnia, who meet threshold scores on one or more self-reported inventories for the same. This includes the Insomnia Severity Index (ISI, ≥ 8), the Perceived Stress Index (PSS, ≥ 14), or the Generalized Anxiety Disorder 7-item (GAD-7, ≥ 5) scale.

Exclusion Criteria:

* Unable, unwilling, or incompetent to provide informed consent/assent.
* Physically unable to come to the study visits, or to sit comfortably in a chair for up to 1.5 hours.
* Severe hearing impairment (because the subject will be using ear buds during CR).
* Weight is over the chair limit (285 pounds).
* Currently in another active intervention research study.
* Prior use of HIRREM, Brainwave Optimization, Cereset, or a wearable configuration of the same (B2, or B2v2) within the last 3 years.
* Prior use of electroconvulsive therapy (ECT).
* Prior use of transcranial magnetic stimulation (TMS), transcranial direct current stimulation (TDCS), alpha stimulation, neurofeedback, biofeedback, or deep brain stimulation (DBS) within one month before enrollment.
* Known seizure disorder.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate Variability | Baseline, and V3 (4-6 weeks after V2)
  Heart rate variability is measured in the time domain as standard deviation of beat-to-beat interval (SDNN, milliseconds). For calculation of SDNN, the R-R intervals are visually inspected, and data considered as artifact is manually removed. Heart rate are acquired from 10 minute recordings of noninvasive finger arterial pressure measurements and ECG with participants lying quietly, supine. Systolic BP and beat to beat, RR intervals files generated via the data acquisition system (BIOPAC acquisition system and Acknowledge 4.2 software, Santa Barbara, CA), at 1000 Hz, are analyzed using Nevrokard BRS software (Nevrokard BRS, Medistar, Ljubljana, Slovenia). Analysis is conducted on the first complete 5-minute epoch that is considered to be acceptable for analysis.
Change in Baroreflex Sensitivity | Baseline, and V3 (4-6 weeks after V2)
  BRS calculated by this method is based on quantification of sequences of at least three beats (n) in which SBP consecutively increases (UP sequence) or decreases (DOWN sequence), which are accompanied by changes in the same direction of the RRI of subsequent beats (n+1). The software scans the RRI and SBP records, identifies sequences, and calculates linear correlation between RRI and SBP for each sequence. The mean of all individual regression coefficients (slopes), a measure of sequence BRS, is calculated for Sequence UP, DOWN and ALL (ms/mmHg). Blood pressure and heart rate are acquired from 10 minute recordings of noninvasive finger arterial pressure measurements and ECG with participants lying quietly, supine. Systolic BP and beat to beat, RR intervals files generated via the data acquisition system (BIOPAC acquisition system and Acknowledge 4.2 software, Santa Barbara, CA), at 1000 Hz, are analyzed using Nevrokard BRS software (Nevrokard BRS, Medistar, Ljubljana, Slovenia).
Change in Blood Pressure Variability | Baseline, and V3 (4-6 weeks after V2)
  Systolic BP and beat to beat, RR intervals (RRI) files generated via the data acquisition system (BIOPAC acquisition system and software, Santa Barbara, CA) at 1000 Hz are analyzed using Nevrokard SA-BRS software (by Nevrokard Kiauta, d.o.o., Izola, Slovenia) for measures BPV.Frequency Method. Power spectral densities of SBP and RRI oscillations are computed by 512 points Fast Fourier Transform (FFT) and integrated over specified frequency ranges (LF: 0.04-0.15 Hz; HF: 0.15-0.4 Hz).

SECONDARY OUTCOMES:
Change in Insomnia Severity Index (ISI) | Baseline, V2 (0-14 days after final session), and V3 (4-6 weeks after V2)
  The severity of insomnia symptoms is measured using the ISI with each data collection visit. The ISI is a 7 question measure, with responses from 0-4 for each question, yielding scores ranging from 0-28. Higher scores indicate the strength of the insomnia severity.
Change in Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline, V2 (0-14 days after final session), and V3 (4-6 weeks after V2)
  The CES-D is a 20-item survey assessing affective depressive symptomatology to screen for risk of depression. Scores range from 0-60, with a score of 16 commonly used as a clinically relevant cut-off. Higher scores indicate the presence of more symptomatology.
Change in Generalized Anxiety Disorder-7 (GAD-7) | Baseline, V2 (0-14 days after final session), and V3 (4-6 weeks after V2)
  The GAD-7 is a seven item screening tool for anxiety that is widely used in primary care. Scores range from 0-21. A lower score denotes a lower level of anxiety.
Change in Perceived Stress Scale (PSS) | Baseline, V2 (0-14 days after final session), and V3 (4-6 weeks after V2)
  The PSS is a ten-item psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Scores range from 0-40. A lower score denotes a lower level of perceived stress.

OTHER OUTCOMES:
Change in Quality of Life Scale (QOLS) | Baseline, V2 (0-14 days after final session), and V3 (4-6 weeks after V2)
  The QOLS is a 16-item scale that was modified from a 15-item scale used in chronic disease patients. Topics include different components of daily life such as relationships, community engagement, personal fulfillment, and recreation. Each item is scaled from 1 to 7 and a sum score is calculated to represent higher levels of satisfaction in life (range is 16-112).
Change in PTSD Checklist for Civilians (PCL-C) | Baseline, V2 (0-14 days after final session), and V3 (4-6 weeks after V2)
  The PCL-C measures the American Psychiatric Association's Diagnostic and statistical manual of mental disorders (DSM-IV) Criteria B, C, & D of PTSD symptoms based on traumatic life experience related to civilians. Seventeen items are rated on a Likert scale with a composite score range of 17 to 85. A score of 44 or higher correlates with probability of civilian-related PTSD.
Change in Blood Pressure | Baseline, and V3 (4-6 weeks after V2)
  BP measurements will be obtained using an automate oscillometric blood pressure device. Three samples will be obtained and the last two averaged to get the value that will be used as the reading for that visit.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Tegeler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Scienc\ess, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hale TS, Smalley SL, Walshaw PD, Hanada G, Macion J, McCracken JT, McGough JJ, Loo SK. Atypical EEG beta asymmetry in adults with ADHD. Neuropsychologia. 2010 Oct;48(12):3532-9. doi: 10.1016/j.neuropsychologia.2010.08.002. Epub 2010 Aug 10. PMID 20705076
- [Background] Hale TS, Smalley SL, Dang J, Hanada G, Macion J, McCracken JT, McGough JJ, Loo SK. ADHD familial loading and abnormal EEG alpha asymmetry in children with ADHD. J Psychiatr Res. 2010 Jul;44(9):605-15. doi: 10.1016/j.jpsychires.2009.11.012. Epub 2009 Dec 16. PMID 20006344
- [Background] Hale TS, Smalley SL, Hanada G, Macion J, McCracken JT, McGough JJ, Loo SK. Atypical alpha asymmetry in adults with ADHD. Neuropsychologia. 2009 Aug;47(10):2082-8. doi: 10.1016/j.neuropsychologia.2009.03.021. Epub 2009 Apr 5. PMID 19467358
- [Background] Lazarev VV, Pontes A, Mitrofanov AA, deAzevedo LC. Interhemispheric asymmetry in EEG photic driving coherence in childhood autism. Clin Neurophysiol. 2010 Feb;121(2):145-52. doi: 10.1016/j.clinph.2009.10.010. Epub 2009 Dec 1. PMID 19951847
- [Background] Stroganova TA, Nygren G, Tsetlin MM, Posikera IN, Gillberg C, Elam M, Orekhova EV. Abnormal EEG lateralization in boys with autism. Clin Neurophysiol. 2007 Aug;118(8):1842-54. doi: 10.1016/j.clinph.2007.05.005. Epub 2007 Jun 19. PMID 17581774
- [Background] Thibodeau R, Jorgensen RS, Kim S. Depression, anxiety, and resting frontal EEG asymmetry: a meta-analytic review. J Abnorm Psychol. 2006 Nov;115(4):715-29. doi: 10.1037/0021-843X.115.4.715. PMID 17100529
- [Background] Avram J, Baltes FR, Miclea M, Miu AC. Frontal EEG activation asymmetry reflects cognitive biases in anxiety: evidence from an emotional face Stroop task. Appl Psychophysiol Biofeedback. 2010 Dec;35(4):285-92. doi: 10.1007/s10484-010-9138-6. PMID 20607389
- [Background] Spironelli C, Penolazzi B, Angrilli A. Dysfunctional hemispheric asymmetry of theta and beta EEG activity during linguistic tasks in developmental dyslexia. Biol Psychol. 2008 Feb;77(2):123-31. doi: 10.1016/j.biopsycho.2007.09.009. Epub 2007 Oct 2. PMID 17997211
- [Background] Moscovitch DA, Santesso DL, Miskovic V, McCabe RE, Antony MM, Schmidt LA. Frontal EEG asymmetry and symptom response to cognitive behavioral therapy in patients with social anxiety disorder. Biol Psychol. 2011 Jul;87(3):379-85. doi: 10.1016/j.biopsycho.2011.04.009. Epub 2011 May 13. PMID 21571033
- [Background] Kemp AH, Griffiths K, Felmingham KL, Shankman SA, Drinkenburg W, Arns M, Clark CR, Bryant RA. Disorder specificity despite comorbidity: resting EEG alpha asymmetry in major depressive disorder and post-traumatic stress disorder. Biol Psychol. 2010 Oct;85(2):350-4. doi: 10.1016/j.biopsycho.2010.08.001. Epub 2010 Aug 11. PMID 20708650
- [Background] Rabe S, Beauducel A, Zollner T, Maercker A, Karl A. Regional brain electrical activity in posttraumatic stress disorder after motor vehicle accident. J Abnorm Psychol. 2006 Nov;115(4):687-98. doi: 10.1037/0021-843X.115.4.687. PMID 17100526
- [Background] Metzger LJ, Paige SR, Carson MA, Lasko NB, Paulus LA, Pitman RK, Orr SP. PTSD arousal and depression symptoms associated with increased right-sided parietal EEG asymmetry. J Abnorm Psychol. 2004 May;113(2):324-9. doi: 10.1037/0021-843X.113.2.324. PMID 15122952
- [Background] Marzano C, Ferrara M, Sforza E, De Gennaro L. Quantitative electroencephalogram (EEG) in insomnia: a new window on pathophysiological mechanisms. Curr Pharm Des. 2008;14(32):3446-55. doi: 10.2174/138161208786549326. PMID 19075720
- [Background] Wolynczyk-Gmaj D, Szelenberger W. Waking EEG in primary insomnia. Acta Neurobiol Exp (Wars). 2011;71(3):387-92. doi: 10.55782/ane-2011-1860. PMID 22068747
- [Background] Riemann D, Spiegelhalder K, Feige B, Voderholzer U, Berger M, Perlis M, Nissen C. The hyperarousal model of insomnia: a review of the concept and its evidence. Sleep Med Rev. 2010 Feb;14(1):19-31. doi: 10.1016/j.smrv.2009.04.002. Epub 2009 May 28. PMID 19481481
- [Background] Cohen H, Benjamin J, Geva AB, Matar MA, Kaplan Z, Kotler M. Autonomic dysregulation in panic disorder and in post-traumatic stress disorder: application of power spectrum analysis of heart rate variability at rest and in response to recollection of trauma or panic attacks. Psychiatry Res. 2000 Sep 25;96(1):1-13. doi: 10.1016/s0165-1781(00)00195-5. PMID 10980322
- [Background] Katz-Leurer M, Rotem H, Keren O, Meyer S. Heart rate and heart rate variability at rest and during exercise in boys who suffered a severe traumatic brain injury and typically-developed controls. Brain Inj. 2010 Feb;24(2):110-4. doi: 10.3109/02699050903508234. PMID 20085448
- [Background] Beckham JC, Taft CT, Vrana SR, Feldman ME, Barefoot JC, Moore SD, Mozley SL, Butterfield MI, Calhoun PS. Ambulatory monitoring and physical health report in Vietnam veterans with and without chronic posttraumatic stress disorder. J Trauma Stress. 2003 Aug;16(4):329-35. doi: 10.1023/A:1024457700599. PMID 12895015
- [Background] Spiegelhalder K, Fuchs L, Ladwig J, Kyle SD, Nissen C, Voderholzer U, Feige B, Riemann D. Heart rate and heart rate variability in subjectively reported insomnia. J Sleep Res. 2011 Mar;20(1 Pt 2):137-45. doi: 10.1111/j.1365-2869.2010.00863.x. PMID 20626615
- [Background] Tobaldini E, Nobili L, Strada S, Casali KR, Braghiroli A, Montano N. Heart rate variability in normal and pathological sleep. Front Physiol. 2013 Oct 16;4:294. doi: 10.3389/fphys.2013.00294. PMID 24137133
- [Background] Tsuji H, Larson MG, Venditti FJ Jr, Manders ES, Evans JC, Feldman CL, Levy D. Impact of reduced heart rate variability on risk for cardiac events. The Framingham Heart Study. Circulation. 1996 Dec 1;94(11):2850-5. doi: 10.1161/01.cir.94.11.2850. PMID 8941112
- [Background] Dekker JM, Schouten EG, Klootwijk P, Pool J, Swenne CA, Kromhout D. Heart rate variability from short electrocardiographic recordings predicts mortality from all causes in middle-aged and elderly men. The Zutphen Study. Am J Epidemiol. 1997 May 15;145(10):899-908. doi: 10.1093/oxfordjournals.aje.a009049. PMID 9149661
- [Background] Beauchaine TP, Thayer JF. Heart rate variability as a transdiagnostic biomarker of psychopathology. Int J Psychophysiol. 2015 Nov;98(2 Pt 2):338-350. doi: 10.1016/j.ijpsycho.2015.08.004. Epub 2015 Aug 11. PMID 26272488
- [Background] Lee EA, Bissett JK, Carter MA, Cowan PA, Pyne JM, Speck PM, Theus SA, Tolley EA. Preliminary findings of the relationship of lower heart rate variability with military sexual trauma and presumed posttraumatic stress disorder. J Trauma Stress. 2013 Apr;26(2):249-56. doi: 10.1002/jts.21797. PMID 23568414
- [Background] Shah AJ, Lampert R, Goldberg J, Veledar E, Bremner JD, Vaccarino V. Posttraumatic stress disorder and impaired autonomic modulation in male twins. Biol Psychiatry. 2013 Jun 1;73(11):1103-10. doi: 10.1016/j.biopsych.2013.01.019. Epub 2013 Feb 21. PMID 23434412
- [Background] Minassian A, Geyer MA, Baker DG, Nievergelt CM, O'Connor DT, Risbrough VB; Marine Resiliency Study Team. Heart rate variability characteristics in a large group of active-duty marines and relationship to posttraumatic stress. Psychosom Med. 2014 May;76(4):292-301. doi: 10.1097/PSY.0000000000000056. PMID 24804881
- [Background] Park J, Marvar PJ, Liao P, Kankam ML, Norrholm SD, Downey RM, McCullough SA, Le NA, Rothbaum BO. Baroreflex dysfunction and augmented sympathetic nerve responses during mental stress in veterans with post-traumatic stress disorder. J Physiol. 2017 Jul 15;595(14):4893-4908. doi: 10.1113/JP274269. Epub 2017 Jun 14. PMID 28503726
- [Background] Park JE, Lee JY, Kang SH, Choi JH, Kim TY, So HS, Yoon IY. Heart rate variability of chronic posttraumatic stress disorder in the Korean veterans. Psychiatry Res. 2017 Sep;255:72-77. doi: 10.1016/j.psychres.2017.05.011. Epub 2017 May 9. PMID 28528244
- [Background] Minassian A, Maihofer AX, Baker DG, Nievergelt CM, Geyer MA, Risbrough VB; Marine Resiliency Study Team. Association of Predeployment Heart Rate Variability With Risk of Postdeployment Posttraumatic Stress Disorder in Active-Duty Marines. JAMA Psychiatry. 2015 Oct;72(10):979-86. doi: 10.1001/jamapsychiatry.2015.0922. PMID 26353072
- [Background] Pyne JM, Constans JI, Wiederhold MD, Gibson DP, Kimbrell T, Kramer TL, Pitcock JA, Han X, Williams DK, Chartrand D, Gevirtz RN, Spira J, Wiederhold BK, McCraty R, McCune TR. Heart rate variability: Pre-deployment predictor of post-deployment PTSD symptoms. Biol Psychol. 2016 Dec;121(Pt A):91-98. doi: 10.1016/j.biopsycho.2016.10.008. Epub 2016 Oct 20. PMID 27773678
- [Background] Kleiger RE, Miller JP, Bigger JT Jr, Moss AJ. Decreased heart rate variability and its association with increased mortality after acute myocardial infarction. Am J Cardiol. 1987 Feb 1;59(4):256-62. doi: 10.1016/0002-9149(87)90795-8. PMID 3812275
- [Background] Carnethon MR, Golden SH, Folsom AR, Haskell W, Liao D. Prospective investigation of autonomic nervous system function and the development of type 2 diabetes: the Atherosclerosis Risk In Communities study, 1987-1998. Circulation. 2003 May 6;107(17):2190-5. doi: 10.1161/01.CIR.0000066324.74807.95. Epub 2003 Apr 14. PMID 12695289
- [Background] Chandra P, Sands RL, Gillespie BW, Levin NW, Kotanko P, Kiser M, Finkelstein F, Hinderliter A, Pop-Busui R, Rajagopalan S, Saran R. Predictors of heart rate variability and its prognostic significance in chronic kidney disease. Nephrol Dial Transplant. 2012 Feb;27(2):700-9. doi: 10.1093/ndt/gfr340. Epub 2011 Sep 12. PMID 21765187
- [Background] Marsac J. [Heart rate variability: a cardiometabolic risk marker with public health implications]. Bull Acad Natl Med. 2013 Jan;197(1):175-86. French. PMID 24672989
- [Background] Thayer JF, Hansen AL, Saus-Rose E, Johnsen BH. Heart rate variability, prefrontal neural function, and cognitive performance: the neurovisceral integration perspective on self-regulation, adaptation, and health. Ann Behav Med. 2009 Apr;37(2):141-53. doi: 10.1007/s12160-009-9101-z. Epub 2009 May 8. PMID 19424767
- [Background] Nolan RP, Jong P, Barry-Bianchi SM, Tanaka TH, Floras JS. Effects of drug, biobehavioral and exercise therapies on heart rate variability in coronary artery disease: a systematic review. Eur J Cardiovasc Prev Rehabil. 2008 Aug;15(4):386-96. doi: 10.1097/HJR.0b013e3283030a97. PMID 18677161
- [Background] Lee SW, Gerdes L, Tegeler CL, Shaltout HA, Tegeler CH. A bihemispheric autonomic model for traumatic stress effects on health and behavior. Front Psychol. 2014 Aug 1;5:843. doi: 10.3389/fpsyg.2014.00843. eCollection 2014. PMID 25136325
- [Background] Bellesi M, Riedner BA, Garcia-Molina GN, Cirelli C, Tononi G. Enhancement of sleep slow waves: underlying mechanisms and practical consequences. Front Syst Neurosci. 2014 Oct 28;8:208. doi: 10.3389/fnsys.2014.00208. eCollection 2014. PMID 25389394
- [Background] Gerdes L, Gerdes P, Lee SW, H Tegeler C. HIRREM: a noninvasive, allostatic methodology for relaxation and auto-calibration of neural oscillations. Brain Behav. 2013 Mar;3(2):193-205. doi: 10.1002/brb3.116. Epub 2013 Jan 14. PMID 23532171
- [Background] Sterling P. Allostasis: a model of predictive regulation. Physiol Behav. 2012 Apr 12;106(1):5-15. doi: 10.1016/j.physbeh.2011.06.004. Epub 2011 Jun 12. PMID 21684297
- [Background] Tegeler CH, Kumar SR, Conklin D, Lee SW, Gerdes L, Turner DP, Tegeler CL, C Fidali B, Houle TT. Open label, randomized, crossover pilot trial of high-resolution, relational, resonance-based, electroencephalic mirroring to relieve insomnia. Brain Behav. 2012 Nov;2(6):814-24. doi: 10.1002/brb3.101. Epub 2012 Oct 28. PMID 23170244
- [Background] Tegeler CH, Tegeler CL, Cook JF, Lee SW, Pajewski NM. Reduction in menopause-related symptoms associated with use of a noninvasive neurotechnology for autocalibration of neural oscillations. Menopause. 2015 Jun;22(6):650-5. doi: 10.1097/GME.0000000000000422. PMID 25668305
- [Background] Tegeler CH, Tegeler CL, Cook JF, Lee SW, Gerdes L, Shaltout HA, Miles CM, Simpson SL. A Preliminary Study of the Effectiveness of an Allostatic, Closed-Loop, Acoustic Stimulation Neurotechnology in the Treatment of Athletes with Persisting Post-concussion Symptoms. Sports Med Open. 2016 Dec;2(1):39. doi: 10.1186/s40798-016-0063-y. Epub 2016 Sep 14. PMID 27747793
- [Background] Tegeler CL, Gerdes L, Shaltout HA, Cook JF, Simpson SL, Lee SW, Tegeler CH. Successful use of closed-loop allostatic neurotechnology for post-traumatic stress symptoms in military personnel: self-reported and autonomic improvements. Mil Med Res. 2017 Dec 22;4(1):38. doi: 10.1186/s40779-017-0147-0. PMID 29502530
- [Background] Fortunato JE, Tegeler CL, Gerdes L, Lee SW, Pajewski NM, Franco ME, Cook JF, Shaltout HA, Tegeler CH. Use of an allostatic neurotechnology by adolescents with postural orthostatic tachycardia syndrome (POTS) is associated with improvements in heart rate variability and changes in temporal lobe electrical activity. Exp Brain Res. 2016 Mar;234(3):791-8. doi: 10.1007/s00221-015-4499-y. Epub 2015 Dec 8. PMID 26645307
- [Background] Tegeler CH, Shaltout HA, Tegeler CL, Gerdes L, Lee SW. Rightward dominance in temporal high-frequency electrical asymmetry corresponds to higher resting heart rate and lower baroreflex sensitivity in a heterogeneous population. Brain Behav. 2015 Jun;5(6):e00343. doi: 10.1002/brb3.343. Epub 2015 May 1. PMID 26085968
- [Background] Lee SW, Laurienti PJ, Burdette JH, Tegeler CL, Morgan AR, Simpson SL, Gerdes L, Tegeler CH. Functional Brain Network Changes Following Use of an Allostatic, Closed-Loop, Acoustic Stimulation Neurotechnology for Military-Related Traumatic Stress. J Neuroimaging. 2019 Jan;29(1):70-78. doi: 10.1111/jon.12571. Epub 2018 Oct 10. PMID 30302866
- [Background] Tegeler CL, Howard LJ, Schmidt KD, Cook JF, Kumar S, Simpson SL, Lee SW, Gerdes L, Tegeler CH. 0389 USE OF A CLOSED-LOOP ACOUSTIC STIMULATION NEUROTECHNOLOGY IMPROVES SYMPTOMS OF MODERATE TO SEVERE INSOMNIA: RESULTS OF A PLACEBO-CONTROLLED TRIAL. Sleep. 2017;40:A145-A.
- [Background] Shaltout HA, Tegeler CL, Lee SW, Tegeler CH. 0363 IN SUBJECTS WITH INSOMNIA, USE OF A CLOSED-LOOP ACOUSTIC STIMULATION NEUROTECHNOLOGY IMPROVES HEART RATE VARIABILITY AND BAROREFLEX SENSITIVITY: RESULTS OF A PLACEBO-CONTROLLED CLINICAL TRIAL. Sleep. 2017;40:A135-A
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Kaplan NM RB. Technique of blood pressure measurement in the diagnosis of hypertension. UpToDate. Barkris GL, Sheridan AM, eds. Waltham, MA; 2010.
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Radloff LS. The CES-D Scale: A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement. 1977;1:385-401.
- [Background] Smarr KL, Keefer AL. Measures of depression and depressive symptoms: Beck Depression Inventory-II (BDI-II), Center for Epidemiologic Studies Depression Scale (CES-D), Geriatric Depression Scale (GDS), Hospital Anxiety and Depression Scale (HADS), and Patient Health Questionnaire-9 (PHQ-9). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S454-66. doi: 10.1002/acr.20556. No abstract available. PMID 22588766
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] FW W, BT L, DS H, JA H, TM K. The PTSD Checklist (PCL): Reliability, validity, and diagnostic utility. 9th Annual Meeting of the International Society for Traumatic Stress Studies. San Antonio, TX.
- [Background] Blanchard EB, Jones-Alexander J, Buckley TC, Forneris CA. Psychometric properties of the PTSD Checklist (PCL). Behav Res Ther. 1996 Aug;34(8):669-73. doi: 10.1016/0005-7967(96)00033-2. PMID 8870294
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Offenbacher M, Sauer S, Kohls N, Waltz M, Schoeps P. Quality of life in patients with fibromyalgia: validation and psychometric properties of the German Quality of Life Scale (QOLS-G). Rheumatol Int. 2012 Oct;32(10):3243-52. doi: 10.1007/s00296-011-2184-4. Epub 2011 Oct 30. PMID 22038277
- [Background] Burckhardt CS, Anderson KL. The Quality of Life Scale (QOLS): reliability, validity, and utilization. Health Qual Life Outcomes. 2003 Oct 23;1:60. doi: 10.1186/1477-7525-1-60. PMID 14613562
- [Background] Burckhardt CS, Woods SL, Schultz AA, Ziebarth DM. Quality of life of adults with chronic illness: a psychometric study. Res Nurs Health. 1989 Dec;12(6):347-54. doi: 10.1002/nur.4770120604. PMID 2602575
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Background] Eckner JT, Kutcher JS, Richardson JK. Pilot evaluation of a novel clinical test of reaction time in national collegiate athletic association division I football players. J Athl Train. 2010 Jul-Aug;45(4):327-32. doi: 10.4085/1062-6050-45.4.327. PMID 20617905
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Bradley KA, Bush KR, Epler AJ, Dobie DJ, Davis TM, Sporleder JL, Maynard C, Burman ML, Kivlahan DR. Two brief alcohol-screening tests From the Alcohol Use Disorders Identification Test (AUDIT): validation in a female Veterans Affairs patient population. Arch Intern Med. 2003 Apr 14;163(7):821-9. doi: 10.1001/archinte.163.7.821. PMID 12695273
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] Bradley KA, DeBenedetti AF, Volk RJ, Williams EC, Frank D, Kivlahan DR. AUDIT-C as a brief screen for alcohol misuse in primary care. Alcohol Clin Exp Res. 2007 Jul;31(7):1208-17. doi: 10.1111/j.1530-0277.2007.00403.x. Epub 2007 Apr 19. PMID 17451397